CLINICAL TRIAL: NCT00003364
Title: A Randomised Study of Timing of Thoracic Irradiation in Small Cell Lung Cancer (Study 8)
Brief Title: Radiation Therapy Plus Combination Chemotherapy In Treating Patients With Limited Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Lung Cancer Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066349; LLCG-TR8SCLC; EU-98011
Record Dates: First submitted 1999-11-01; First posted 2004-01-23 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-05

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Cyclophosphamide; Doxorubicin; Etoposide; Vincristine; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug with radiation therapy may kill more tumor cells. The best timing for radiation therapy and combination chemotherapy in treating limited stage small cell lung cancer is not yet known .

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy given at different times along with combination chemotherapy in treating patients with limited stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether long term survival is affected by the timing of thoracic radiotherapy in patients with limited stage small cell lung cancer who are receiving combination chemotherapy. II. Determine whether the development of local recurrence and distant metastases are affected by the timing of thoracic radiotherapy in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by center. All patients receive cyclophosphamide, doxorubicin, and vincristine by IV bolus alternating with 3 days of daily etoposide IV infusion over 60-120 minutes and cisplatin IV infusion over 30 minutes. This treatment alternates every 3 weeks for six courses. Patients are randomized to have thoracic radiotherapy either with course 2 (arm I) or with course 6 (arm II) of chemotherapy. Patients in arm I are given 1 week of rest between radiotherapy and the second course of chemotherapy. If there is no disease progression after chemotherapy and locoregional irradiation, and a repeat brain scan is negative, patients receive prophylactic brain irradiation. Patients are followed monthly for the first year and then every 2 months thereafter.

PROJECTED ACCRUAL: This study will accrue 398 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed limited stage small cell lung cancer Limited disease defined as within the hemithorax, mediastinum, or ipsilateral supraclavicular nodes No evidence of extensive disease (i.e., contralateral lung or contralateral supraclavicular nodes) No metastatic disease Measurable or evaluable disease

PATIENT CHARACTERISTICS: Age: Under 75 Performance status: ECOG 0-3 Life expectancy: At least 8 weeks Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 mg/dL Renal: Creatinine normal OR Creatinine clearance greater than 50 mL/min OR Pentetic acid/ethylenediaminetetraacetic acid clearance greater than 70 mL/min Cardiovascular: No myocardial infarction in the 3 months prior to diagnosis No pericardial effusion Pulmonary: No pleural effusion seen on chest x-ray Pleural effusion identified on CT allowed, if not visible on chest x-ray Other: No medical condition that excludes the use of chemotherapy or thoracic irradiation Must be able to tolerate the prescribed study radiotherapy No other malignant tumor for at least 3 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy No concurrent chemotherapy Endocrine therapy: Concurrent prednisone or other corticosteroids for hypercalcemia allowed Radiotherapy: No prior radiotherapy Surgery: Not specified

Max Age: 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 1993-01; Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen G. Spiro, Study Chair — University College London Hospitals
Locations (14):
- United Kingdom (14):
  - Heatherwood Hospital, Ascot, England
  - Royal Sussex County Hospital, Brighton, England
  - Addenbrooke's NHS Trust, Cambridge, England
  - Broomfield Hospital, Chelmsford, Essex, England
  - Essex County Hospital, Colchester, England
  - Royal Free Hospital, Hampstead, London, England
  - Cookridge Hospital, Leeds, England
  - Saint Bartholomew's Hospital, London, England
  - Guy's and St. Thomas' Hospitals Trust, London, England
  - Charing Cross Hospital, London, England
  - Middlesex Hospital- Meyerstein Institute, London, England
  - Mount Vernon Hospital, Northwood, England
  - Peterborough Hospitals Trust, Peterborough, England
  - Southend NHS Trust Hospital, Westcliff-on-Sea, England

REFERENCES:
- [Result] Spiro SG, James LE, Rudd RM, Trask CW, Tobias JS, Snee M, Gilligan D, Murray PA, Ruiz de Elvira MC, O'Donnell KM, Gower NH, Harper PG, Hackshaw AK; London Lung Cancer Group. Early compared with late radiotherapy in combined modality treatment for limited disease small-cell lung cancer: a London Lung Cancer Group multicenter randomized clinical trial and meta-analysis. J Clin Oncol. 2006 Aug 20;24(24):3823-30. doi: 10.1200/JCO.2005.05.3181. PMID 16921033